CLINICAL TRIAL: NCT06581575
Title: A Phase 2, Randomized, Triple-Blinded, Active-Controlled Study to Assess the Safety and Immunogenicity of an Investigational Herpes Zoster (HZ) Vaccine, JCXH-105, in Healthy Subjects ≥ 50 Years of Age
Brief Title: A Phase 2 Study to Evaluate JCXH-105, an srRNA-based Herpes Zoster Vaccine
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Immorna Biotherapeutics, Inc. (Industry)
Collaborators: Tigermed Consulting Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: JCXH-105-021
Record Dates: First submitted 2024-08-29; First posted 2024-09-03 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Herpes Zoster (HZ); Infectious Diseases; Shingles
Keywords: srRNA; Herpes Zoster (HZ) vaccination; Healthy Subjects
MeSH Terms: conditions — Herpes Zoster; Communicable Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Triple-blinded study
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Investigational Product (Experimental): Participants randomized to this arm will be given the investigational product (JCXH-105).
  Interventions: Biological: JCXH-105
- Active Control (Active Comparator): Participants randomized to this arm will be given the FDA approved Shingrix.
  Interventions: Biological: Shingrix

INTERVENTIONS:
Biological: JCXH-105 — IM injection
  Arms: Investigational Product
Biological: Shingrix — IM injection
  Arms: Active Control

SUMMARY:
The goal of this clinical trial is to assess the safety and immunogenicity of an srRNA-based vaccine, JCXH-105, in the prevention of Herpes Zoster (Shingles).

Subjects will be randomized to receive either JCXH-105 or Shingrix.

DETAILED DESCRIPTION:
This Phase 2 study plans to enroll a total of 460 subjects.

This will be an active-controlled study in healthy male and/or female subjects 50 years of age or older. Subjects will be randomized 1:1 to receive either JCXH-105 or Shingrix. The study vaccine will be administered in two doses approximately 2 months apart. The subject will receive a single intramuscular (IM) injection of JCXH-105 or Shingrix on Day 1 (Dose 1) and again on Day 61 ± 7 days (Dose 2). For each subject, Dose 1 and Dose 2 are the same study vaccine based on randomization on Day 1. A total of 460 subjects will be enrolled into this trial and vaccinated with either JCXH-105 (n=230) or Shingrix (n=230).

ELIGIBILITY:
Key Inclusion Criteria:

* Sex: Male or female; female subjects may be of childbearing potential, of nonchildbearing potential, or postmenopausal.
* Age: ≥ 50 years of age at screening.
* Status: Healthy subjects.
* Subjects must agree to not be vaccinated with any HZ vaccine while participating in this study.
* Subjects must agree to not be vaccinated with any RNA-based vaccines (e.g., Spikevax, Comirnaty, etc.) 30 days before Dose 1 through 30 days after Dose 2 (a 4-month period).

Key Exclusion Criteria:

* Subjects with a history of HZ within the past 10 years or current diagnosis of HZ.
* Previous vaccination against HZ.
* Subjects with any respiratory illness deemed clinically relevant by the Investigator within the past month OR hospitalization >24 hours for any reason within the past month prior to the first vaccine administration (JCXH-105 or Shingrix).
* Subjects who are acutely ill or febrile with body temperature ≥ 38.0º Celsius/100.4º Fahrenheit 72 hours prior to or at the Screening visit or on Day 1 pre-dose. Subjects meeting this criterion may be rescheduled within an allowable window with approval from the Sponsor.
* Subjects with history or current diagnosis of congenital or acquired immunodeficiency/immunocompromising/immunosuppressive conditions, asplenia, or recurrent severe infections. Certain immune-mediated conditions (e.g., Hashimoto thyroiditis) that are well controlled and stable are allowed.
* Subjects with history of myocarditis or pericarditis, or with AEs (including anaphylaxis and severe hypersensitivity) after mRNA vaccination that are in nature and severity beyond the common expected AEs and necessitating medical intervention.
* Subjects who received any non-live vaccine within 14 days prior to Day 1 (first dose of JCXH-105 or Shingrix).
* Subjects who received within 28 days prior to Day 1 (first dose of JCXH-105 or Shingrix): (1) Any live vaccine, (2) Immunomodulators or immune-suppressive medication, (3) Granulocyte or granulocyte-macrophage colony-stimulating factor, (4) Three or more consecutive days of systemic corticosteroids. Note: subjects on stable-dose steroid replacement (for chronic disease such as iatrogenic deficiency) of prednisone ≤10 mg/day or equivalent are allowed and (5) Other investigational agents or devices.
* Subjects receiving systemic antiviral therapy.
* Subjects with a positive screening test for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies, anti-human HIV-1 and 2 antibodies, or syphilis.
* Subjects with a positive screening test for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 467 (Actual)
Dates: Start 2024-10-16 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
SAE Frequency | Day 1 - Day 241 (Week 34)
  Frequency of SAEs characterized by type, severity, duration, and relationship to the vaccine recorded from Day 1 post-vaccine administration through follow-up completion.
Solicited local reaction frequency | Day 1 - Day 7 (After Dose 1), Day 1 - Day 7 (After Dose 2)
  Occurrence of solicited local injection site reactions characterize by frequency, severity, and duration within 7 days after each vaccine administration.
Solicited systemic reaction frequency | Day 1 - Day 7 (After Dose 1), Day 1 - Day 7 (After Dose 2)
  Occurrence of solicited systemic reactions characterize by frequency, severity, and duration within 7 days after each vaccine administration.
AE Frequency | Day 1 - Day 241 (Week 34)
  Adverse events (AEs) including unsolicited AEs and any AEs leading to discontinuation of study vaccine or withdrawal from the study, characterized by frequency, severity, duration, and relationship to the vaccine from Day 1 post-vaccine administration through follow-up completion.
AESIs Frequency | Day 1 - Day 241 (Week 34)
  AESIs characterized by frequency, severity, duration, and relationship to the vaccine from Day 1 post-vaccine administration through follow-up completion.
Medically Attended AE Frequency | Day 1 - Day 241 (Week 34)
  Medically attended AEs (MAAEs) characterized by frequency, severity, duration, and relationship to the vaccine from Day 1 post-vaccine administration through follow-up completion.
Immune-Mediated Adverse Events of Special Interest Frequency | Day 1 - Day 241 (Week 34)
  Immune-mediated adverse events of special interest (imAESIs) characterized by frequency, severity, duration, and relationship to the vaccine (JCXH-105 or Shingrix) recorded from Day 1 post-vaccine administration through follow-up completion.
gE-Specific CD4+ T cell Response Rate | Day 1 - Day 89 (Week 13)
  Response Rate is defined at the percentage of subjects with ≥ 2 folds increase of gE-specific CD4+ T cells expressing 2 or more markers of activation (IFN-γ, IL-2, TNFα, and CD40L) in PBMCs analyzed with flow cytometry with ICS on Day 89 as compared to baseline (Day 1 pre-dose).

SECONDARY OUTCOMES:
Cellular immunogenicity of JCXH-105 | Day 1 - Day 241 (Week 34)
  Frequency of glycoprotein E (gE)-specific CD4+ T cells expressing 2 or more markers of activation (IFN-γ, IL-2, TNF-α, and CD40L) in PBMCs analyzed by flow cytometry with ICS on Day 29, Day 89, and Day 241 as compared to baseline (Day 1 pre-dose).

OTHER OUTCOMES:
Cellular Immunogenicity of JCXH-105 | Day 1 - Day 241 (Week 34)
  Frequency of gE-specific CD8+ T cells expressing 2 or more markers of activation (IFN-γ, IL-2, TNF-α, and CD40L) in PBMCs analyzed by flow cytometry on Day 29, Day 89, and Day 241 as compared to baseline (Day 1 pre-dose).
Humoral immunogenicity of JCXH-105 | Day 1 - Day 241 (Week 34)
  Changes in serum of anti-gE-specific antibody geometric mean titers (GMTs) analyzed with enzyme-linked immunosorbent assay (ELISA) on Day 29, Day 89, and Day 241 as compared to baseline (D1 pre-dose).

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Noble Clinical Research, Tucson, Arizona
  - Long Beach Research Institute, Long Beach, California
  - DM Clinical Research - Chicago, Chicago, Illinois
  - Quality Clinical Research, Omaha, Nebraska
  - DM Clinical Research - New Jersey, Jersey City, New Jersey
  - Delricht Research, Charleston, South Carolina
  - Delricht Research, Prosper, Texas
  - DM Clinical Research - Sugarland, Sugar Land, Texas